CLINICAL TRIAL: NCT02755272
Title: A Randomized Phase II Clinical Trial Assessing the Efficacy and Safety of MK-3475 (Pembrolizumab) in Combination With Carboplatin and Gemcitabine in Patients With Metastatic Triple Negative Breast Cancer
Brief Title: A Study of Pembrolizumab With Carboplatin and Gemcitabine in Patients With Metastatic Triple Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR-076; 16-1013 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Carcinoma Breast Stage IV
Keywords: Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — pembrolizumab; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pembrolizumab with Standard Chemotherapy (Experimental): Pembrolizumab plus standard chemotherapy using carboplatin and gemcitabine.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Gemcitabine
- Standard Chemotherapy Alone (Active Comparator): Standard chemotherapy alone using carboplatin and gemcitabine.
  Interventions: Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Pembrolizumab — IV Infusion of 200 mg given on day one of each 21 day treatment cycle.
  Other Names: MK-3475; Keytruda
  Arms: Pembrolizumab with Standard Chemotherapy
Drug: Carboplatin — IV infusion of a calculated dose (AUC 2 mL/min) given on days one and eight of each 21 day treatment cycle.
  Other Names: Paraplatin
Drug: Gemcitabine — IV infusion of 800 mg/m^2 given on days one and eight of each 21 day treatment cycle.
  Other Names: Gemzar

SUMMARY:
The main purpose of this study is to see if Pembrolizumab in combination with chemotherapy (carboplatin and gemcitabine) is safe and effective in treating patients with metastatic triple negative breast cancer.

Pembrolizumab is a drug which may help the immune system to target and destroy cancer cells. Pembrolizumab has been approved by the FDA for the treatment of advanced melanoma and metastatic non-small cell lung cancer. However, it has not been approved as a treatment for breast cancer.

ELIGIBILITY:
Subject Inclusion Criteria for Part 1: Safety Run-in study

1. Women diagnosed with pathologically confirmed metastatic triple negative invasive breast cancer (centrally confirmed immunophenotype negative for all three receptors ER, PR and HER2).
2. Hormone receptor status (ER and PR) both ≤ 5% by immunohistochemistry, and HER2 status confirmed by means of immunohistochemistry (with 0 or 1+ indicating negative status) or fluorescence in situ hybridization (with amplification ratio < 2.0 indicating negative status).
3. Have either Evaluable disease, or have measurable clinical disease: Measurable disease, defined as at least 1 unidimensionally measurable lesion on a CT scan as defined by RECIST (version v1.1).
4. Age > 18 years.
5. Disease stage: Unresectable metastatic disease.
6. Patients received up to 2 prior regimens for their disease in the metastatic setting.
7. Patients are candidates for chemotherapy with carboplatin and gemcitabine.
8. ECOG performance status 0 - 2.
9. Adequate organ function tests and hematologic indices within 10 days of registration.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female subjects of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
12. Signed written Informed Consent in accordance with regulatory and institutional guidelines

Subject Exclusion Criteria for Part 1: Safety Run-in study

1. Patients participating in another trial of an investigational agent within 4 weeks of the first dose of the study.
2. Patients who received prior therapy using carboplatin/gemcitabine within 12 months prior to enrollment or subjects whose tumor progressed while on treatment with carboplatin or cisplatin.
3. Patients with baseline grade 2 neuropathy.
4. Patients with Hormone-receptor positive breast cancer (ER and/or PR > 5%), and with HER-2 positive breast cancer (by means of immunohistochemistry with 3+ indicating positive status or fluorescence in situ hybridization with amplification ratio ≥2.0 indicating positive status).
5. Diagnosis of immunosuppression or receiving steroid therapy or other immunosuppressive therapy within 4 weeks of the study.
6. Active autoimmune disease or a documented history of autoimmune disease, or a syndrome that has required systemic treatment in the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thryoxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc) is not considered a form of systemic treatment. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects who require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjögren's syndrome will not be excluded from the study.
7. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
8. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
9. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
10. If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
11. Known additional malignancy that progressed and/or required treatment in the last 5 years. Except that for basal and squamous cell carcinoma of the skin or in situ cervical carcinoma that has completed potentially curative therapy.
12. Life expectancy of less than 3 months.
13. Patients known to be carriers of Human Immunodeficiency Virus (HIV1/2).
14. Patients known to be carriers of hepatitis virus B and C.
15. Prior therapy with an anti-programmed cell death 1 (PD-1), anti-programmed cell death 1 ligand (PDL-1), anti-PD-L2, anti-CD137 antibody, or anti-cytotoxic T-lymphocyte -associated antigen-4 (CTLA-4) antibody.
16. Pregnant, breastfeeding, or expecting to conceive children within the projected time of the trial, starting with the pre-screening or screening visit and through 120 days after the last dose of trial treatment.
17. Active infection requiring systemic therapy.
18. Active substance abuse or psychiatric disorders.
19. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
21. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Subject Inclusion Criteria for Part 2 (Randomized Phase II Clinical Trial)

1. Women diagnosed with pathologically confirmed triple negative invasive breast cancer, metastatic (locally confirmed immunophenotype negative for all three receptors ER, PR, HER2).
2. Hormone receptor status (ER and PR) both ≤ 5% by immunohistochemistry, and HER2 status confirmed by means of immunohistochemistry (with 0 or 1+ indicating negative status) or fluorescence in situ hybridization (with amplification ratio < 2.0 indicating negative status).
3. Age > 18 years.
4. Disease stage IV, metastatic unresectable disease.
5. Have measurable clinical disease: Measurable disease, defined as at least 1 unidimensionally measurable lesion on a CT scan as defined by RECIST (version v1.1).
6. Patients received up to 3 prior regimens for their metastatic disease. Prior hormone therapy will not be counted towards the line of therapies.
7. Patients are candidates for chemotherapy with carboplatin and gemcitabine.
8. ECOG performance status 0-2.
9. Adequate organ function tests and hematologic indices within 10 days of registration.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
12. Signed written Informed Consent in accordance with regulatory and institutional guidelines.
13. Have provided tissue from a newly obtained biopsy (an archival tissue sample may be substituted if new biopsy cannot be obtained and by discretion of Principal Investigator only) from a local or distant site and agreed to providing a second newly obtained biopsy after completion of 2 cycles of the study drugs.

Subject Exclusion Criteria for Part 2 (Randomized Phase II Clinical Trial)

1. Patients participating in another trial of an investigational agent within 4 weeks of the first dose of the study.
2. Patients with tumors that cannot be measured or clinically followed (i.e. evaluable disease).
3. Patients with metastatic breast cancer who received prior therapy using carboplatin/gemcitabine within 12months prior to their enrollment or subjects whose tumor progressed while on treatment with carboplatin or cisplatin.
4. Patients with baseline grade 2 neuropathy.
5. Patients with Hormone-receptor positive breast cancer (ER and/or PR > 5%), and with HER-2 positive breast cancer (by means of immunohistochemistry with 3+ indicating positive status or fluorescence in situ hybridization with amplification ratio ≥2.0 indicating positive status).
6. Diagnosis of immunosuppression or receiving steroid therapy or other immunosuppressive therapy within 4 weeks of the study.
7. Active autoimmune disease or a documented history of autoimmune disease, or a syndrome that has required systemic treatment in the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thryoxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc) is not considered a form of systemic treatment. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects who require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjögren's syndrome will not be excluded from the study.
8. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
9. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
10. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
11. If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
12. Known additional malignancy that progressed and/or required treatment in the last 5 years. Except that for basal and squamous cell carcinoma of the skin or in situ cervical carcinoma that has completed potentially curative therapy.
13. Life expectancy of less than 3 months.
14. Patients known to be carriers of Human Immunodeficiency Virus (HIV1/2).
15. Patients known to be carriers of hepatitis virus B and C .
16. Prior therapy with an anti-programmed cell death 1 (PD-1), anti-programmed cell death 1 ligand (PDL-1), anti-PD-L2, anti-CD137 antibody, or anti-cytotoxic T-lymphocyte -associated antigen-4 (CTLA-4) antibody.
17. Pregnant, breastfeeding, or expecting to conceive children within the projected time of the trial, starting with the pre-screening or screening visit and through 120 days after the last dose of trial treatment.
18. Active infection requiring systemic therapy.
19. Active substance abuse or psychiatric disorders.
20. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
21. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
22. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
23. Subjects who do not consent to providing pre and post treatment tissue sample for future research would not be eligible to participate in the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 87 (Estimated)
Dates: Start 2016-05-31 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 24 months
  Evaluate antitumor activity by assessing the percentage of patients with evidence of complete response or partial response per RECIST 1.1 criteria.
Incidence of Treatment-Related Adverse Events | From the first dose of study treatment until 30 days after discontinuation of study treatment.
  The safety and tolerability of Pembrolizumab in Combination with Carboplatin and Gemcitabine will be evaluated from the results of reported signs and symptoms, scheduled physical examinations, vital sign measurements, and clinical laboratory test results.

SECONDARY OUTCOMES:
Clinical Benefit Rate | Up to 24 months
  Evaluate antitumor activity by assessing the percentage of patients with evidence of complete response, partial response, or stable disease per RECIST 1.1 criteria
Progression Free Survival | From the start of treatment until progressive disease or date of death, whichever occurs first (assessed up to 60 months.)
  Evaluate antitumor activity by assessing the time interval from initiation of study drug until progressive disease or death whichever occurs first.
Overall Survival | From the start of treatment until death (assessed up to 60 months.)
  Evaluation of the overall survival rate of patients

OTHER OUTCOMES:
Assessment of Association of PD-L1 Expression with Clinical Benefit Rate | Up to 24 months
Assessment of Association of PD-L1 Expression with Progression Free Survival | Up to 24 months
Assessment of Association of PD-L1 Expression with Overall Survival | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Elias Obeid, MD, Principal Investigator — Fox Chase Cancer Center
Locations (6):
- United States (6):
  - Indiana University, Indianapolis, Indiana
  - Washington University in St. Louis, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin